CLINICAL TRIAL: NCT02305407
Title: Neurocognitive and Radiological Assessments in Adult Patients With Moyamoya Disease Undergoing Surgical Revascularization
Brief Title: Neurocognitive and Radiological Assessments in Adult Moyamoya Undergoing Surgery
Acronym: NRAAMUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yu Lei, MD, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCI2014
Record Dates: First submitted 2014-11-19; First posted 2014-12-02 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgical revascularization (Experimental): Patients will be assigned to either surgical or conservative treatment depending on their clinical symptoms and radiological assessment.
  Interventions: Procedure: Surgical Revascularization
- conservative treatment (Experimental): Normal conservative treatment without surgical intervention.
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Procedure: Surgical Revascularization — Most patients in this group will be performed combined procedures of superficial temporal to middle cerebral artery bypass (STA-MCA) and encephalo-duro-myo-synangiosis (EDMS). Patients not suitable for combined procedures will be performed EDMS.
  Arms: surgical revascularization
Other: Conservative treatment — Patients will be medically treated with antiplatelets, antiepileptics, antihypertensives and vasodilators depending on the presentation.
  Arms: conservative treatment

SUMMARY:
Adult patients with moyamoya disease (MMD) are reported to suffer from considerable impairment of executive function/attention. Although reduced cerebrovascular reserve (CVR) in frontal areas has been detected by perfusion MRI and then confirmed to be associated with executive dysfunction in adult MMD, the structural and functional changes is still unclear with progression of executive dysfunction. Furthermore, it is very important to study the association between the neurocognitive and radiological improvement after surgical revascularization, so as to help detecting cerebral regions which are involved in executive deterioration or improvement after surgery. Then the investigators can determine whether these regions can be used as indicators to decide rational therapeutic schedule and timing of adult MMD with executive dysfunction.

Thus the aim of this study is to primarily find out the neuropsychological and radiological correlates in adult MMD, and then to quantitatively evaluate the effectiveness of surgical revascularization in prevention of executive dysfunction in adult MMD.

DETAILED DESCRIPTION:
Previous studies of adult moyamoya disease (MMD) have revealed that vascular cognitive impairment (VCI) is the consequence of ischemic damage to dynamic factors such as cerebral hypoperfusion, rather than to cerebral gray matter. However, it is still unclear which regions are affected by MMD and how these regions respond to the progressive cognitive decline. In other way, the investigators need to detect spatial patterns in the brain activity of MMD in order to understand its pathophysiological nature.

Surgical revascularization has been accepted as the only effective form of treatment in preventing future ischemic episodes. However, its effectiveness in cognitive protection is still unknown. Thus, the investigators determine to quantitatively evaluate cognitive and radiological outcomes in adult MMD postoperatively and during follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed Chinese people aged over 18 years
* No evidence of recent or remote infarct in the cerebral cortical, basal ganglia, brainstem or cerebellum
* No evidence of recent or remote intracerebral hemorrhage
* Diagnosis confirmed by digital subtraction angiography (DSA) according to Suzuki scale
* No surgical intervention before recruitment
* Physically capable of cognitive testing
* Geographically accessible and reliable for follow-up.

Exclusion Criteria:

* Significant neurological diseases or psychiatric disorders that could affect cognition
* Other cerebrovascular diseases (such as atherosclerosis or vasculitides) likely to cause focal cerebral ischemia
* Concomitant cerebrovascular diseases (such as aneurysms or arteriovenous malformation) that need surgical intervention
* Severe systemic diseases
* Pregnant or perinatal stage women
* Any diseases likely to death within 2 yeas
* Taking drugs such as benzodiazepine clonazepam
* Any contraindications or allergy to aspirin
* Allergy to iodine or radiographic contrast media
* Past history of surgical revascularization
* Concurrent participation in any other experimental treatment trial
* Any condition that in the surgeon's judgment suggests the patient an unsuitable surgical candidate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive outcomes at 3/6/12/24-month follow-up after surgical revascularization or conservative treatment. | 2 years
  Measure neurocognitive outcomes with a battery of neuropsychological tests covering global cognition, executive, memory, language, and visuospatial functions. It involves the Mini-mental state examination (MMSE), the Memory and Executive Screening test (MES), the Trail Making Test (TMT), the Auditory Verbal Learning Test (AVLT), the verbal fluency test (VFT), the Rey-Osterrieth complex figure test (CFT), etc.

SECONDARY OUTCOMES:
The number of participants who suffer from all stroke or death during 30 days to 24 months | 24 months
The number of participants who suffer from all kinds of adverse events related to surgery. | 30 days
Postoperative neurocognitive outcomes before discharge. | average of 1 week after surgery
  Measure neurocognitive outcomes about 1 week after surgery according to participants' physical condition, using the tests mentioned in the primary outcome measurement.
Postoperative radiological outcomes before discharge. | average of 1 week after surgery
  Measure cerebral perfusion simultaneously with neurocognitive testing, using the single photon emission computed tomography (SPECT).
The changes from baseline in modified Rankin scale (mRS) and national institutes of health stroke scale (NIHSS). | at 7 days, 30 days, 3/6/12/24 months
The changes from baseline in single photon emission computed tomography (SPECT). | 2 years
The changes from baseline in blood oxygen level-dependent functional magnetic resonance imaging (BOLD fMRI) during rest. | 2 years
  Data analysis techniques include amplitude of frequency fluctuation (ALFF), regional homogeneity (ReHo), independent component analysis (ICA), voxel-based morphometry analysis (VBM), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiang Gu, MD,PhD, Study Chair — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (1):
- Department of Neurosurgery, Huashan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Su JB, Xi SD, Zhou SY, Zhang X, Jiang SH, Xu B, Chen L, Lei Y, Gao C, Gu YX. Microstructural damage pattern of vascular cognitive impairment: a comparison between moyamoya disease and cerebrovascular atherosclerotic disease. Neural Regen Res. 2019 May;14(5):858-867. doi: 10.4103/1673-5374.249234. PMID 30688272